CLINICAL TRIAL: NCT06766136
Title: The Effect of Education Given to Asthmatic Individuals According to Roy Adaptation Model on Psychosocial Adjustment and Quality of Life
Brief Title: Effectiveness of Asthma Education Program Based on the Roy Adaptation Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Döndü ERDOĞAN İNAN, Lecturer, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: dnd1
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Asthma Patients
Keywords: Asthma patient; Psychosocial Adjustment; Life Quality

STUDY DESIGN:
Intervention Model Description: In this study, stratified sampling based on gender and asthma control test (ACT) was used in this study. [ACT; 24-20, female], [ACT≤19 24-20, female], [ACT; 24-20, male], [ACT≤19 24-20, male] to ensure equal distribution in terms of gender and asthma control test in each group, strata were created. First, a scheme was developed to bi-randomize the gender and asthma control tests so that the experimental and control groups were stratified according to gender and asthma control tests. Permutation was also used to ensure a balance between strata. Block sets were created for each combination of prognostic factors (gender and asthma control test). The experimental and control groups were then randomized into strata using a table of random numbers.
Who Masked: Participant
Masking Description: Single Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma education program (Experimental): Experimental: Asthma education program Experiment group will receive an education program based on Roy Adaptation Model in addition to standard asthma treatment.
  Interventions: Behavioral: Asthma education program
- Standard asthma treatment (No Intervention): No Intervention: Standard asthma treatment

INTERVENTIONS:
Behavioral: Asthma education program — An educational program based on the Roy Adaptation Model in addition to standard asthma treatment.
  Arms: Asthma education program

SUMMARY:
The aim of the study; to determine the effect of the education program given to individuals diagnosed with asthma based on Roy's adjustment model on their psychosocial adjustment to the disease and their quality of life.

DETAILED DESCRIPTION:
In addition to the expected physiological effects of asthma on individuals, the course of the disease and the course of the individual's life will change as the duration of living with the disease increases. In order to improve the attitude towards the disease positively in asthmatic individuals, to ensure asthma control and to improve the quality of life by managing the process well, patients' behaviors against the disease should be improved. Regular repetition of trainings created within the framework of a specific plan to improve adaptation behaviors is one of the recommended steps to empower individuals with chronic diseases during the disease process. In this randomized controlled trial, individuals aged 18-64 years with a diagnosis of asthma, an asthma control test (ACT) score of 24-20 (partial control) or ≤19 (uncontrolled) and no secondary chronic disease other than asthma were included.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-64
* Diagnosed with asthma for at least 6 months
* To live in the city center
* Asthma control test (ACT) score 24-20 (partial control) or ≤19 (uncontrolled)
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* Has a secondary chronic disease other than asthma
* Diagnosed with neuropsychiatric illness
* Individuals with inability to understand or speak Turkish and sensory problems that prevent communication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
"Evaluation of psychosocial adjustment of asthmatic individuals after education with the Psychosocial Adjustment To Illness-Self-Report Scale (PAIS-SR)". | "From enrollment to the end of treatment at 12 weeks"
  Patient Introduction Form This form was prepared by the researcher in line with the literature and consists of 12 questions to determine patient and disease characteristics.
  Psychosocial Adaptation to Illness-Self-Report Scale (PAIS-SR) Psychosocial Adaptation to Illness-Self-Report Scale (PAIS-SR) The Psychosocial Adjustment to Illness - Self-Report Scale was developed by Derogatis in 1986 to assess psychosocial adjustment to illness. The scale consists of 7 sub-dimensions and a total of 46 questions. Scores that can be obtained from the scale vary between "0 - 138". Scores below 35 indicate "good psychosocial adjustment", scores between 35 and 51 indicate moderately "good psychosocial adjustment", and scores above 51 indicate "poor psychosocial adjustment". In the original version of the scale, Cronbach's alpha coefficient was found to be 0.86.

SECONDARY OUTCOMES:
"Evaluation of the quality of life of asthmatic individuals after education with the Asthma Quality of Life Questionnaire (AQLQ)". | "From enrollment to the end of treatment at 12 weeks"
  Patient Introduction Form This form was prepared by the researcher in line with the literature and consists of 12 questions to determine patient and disease characteristics.
  Asthma Quality of Life Questionnaire (AQLQ) The Asthma Quality of Life Questionnaire (AQLQ) is an asthma-specific quality of life scale consisting of 32 questions and 4 subscales developed by Juniper et al. The scale is a 7-point Likert-type scale with "1" representing the lowest and "7" the highest score. The total score of the scale ranges from 32 to 224 and the mean score ranges from 1 to 7. Overall quality of life is calculated by summing and averaging the relevant domain values of all questions and sub-dimensions. An increase in the mean value of the overall and sub-dimensions of the scale increases the quality of life. It was found that the Cronbach alpha coefficients of the sub-dimensions of the scale ranged between 0.81-0.87

CONTACTS AND LOCATIONS:
Overall Officials: Dondu Erdogan Inan, MSc, Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Result] Alpaydin AO, Bora M, Yorgancioglu A, Coskun AS, Celik P. Asthma control test and asthma quality of life questionnaire association in adults. Iran J Allergy Asthma Immunol. 2012 Dec;11(4):301-7. PMID 23264406
- [Result] Ozgen Alpaydin A, Yorgancioglu A, Yilmaz O, Bora M, Goktalay T, Celik P, Yuksel H. Validity and reliability of "Asthma Quality of Life Questionnaire" in a sample of Turkish adult asthmatic patients. Tuberk Toraks. 2011;59(4):321-7. PMID 22233301